CLINICAL TRIAL: NCT06599086
Title: USG-guided Steroid Injection Treatment: Efficacy of in Patients With Bifid Median Nerve Diagnosed Carpal Tunnel Syndrome Versus With Non-bifid Median Nerve Diagnosed Carpal Tunnel Syndrome:A Single-blind Randomized Controlled Study
Brief Title: Efficacy of Steroid Injection in Patients With Bifid Median Nerve Diagnosed Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunus Burak Bayır (Other Government)
Responsible Party: Sponsor-Investigator, Yunus Burak Bayır, Yunus Burak Bayır, Principal İnvestigator, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Perineural steroid Injection
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: corticosteroid; injection; bifid median nerve; carpal tunnel syndrome; variation of median nerve
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Our study was designed as a prospective, double-blind randomized controlled study.Patients who applied to our hospital's PMR outpatient clinic and with moderate carpal tunnel syndrome by EMG will be included in the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The physician performing the evaluation and participants will be blind to which procedure is performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with bifid median nerve diagnosed with carpal tunnel syndrome (Active Comparator): Each patient will receive 2 cc:(1 cc betamethasone dipropionate+1cc saline) perineural injection into the median nerve under US guidance, for 1 session.
  Interventions: Drug: 2 cc:(1 cc betamethasone dipropionate+1cc physiological saline)
- Patients with anatomical variations without median nerve diagnosed with carpal tunnel syndrome (Active Comparator): Each patient will receive 2 cc:(1 cc betamethasone dipropionate+1cc physiological saline) perineural injection into the median nerve under US guidance, for 1 session.
  Interventions: Drug: 2 cc:(1 cc betamethasone dipropionate+1cc physiological saline)

INTERVENTIONS:
Drug: 2 cc:(1 cc betamethasone dipropionate+1cc physiological saline) — Each patient will receive 2 cc:(1 cc betamethasone dipropionate+1cc physiological saline) perineural injection into the median nerve under US guidance, for 1 session.
  Other Names: perineural steroid injection

SUMMARY:
Various median nerve anatomical variations have been reported in the literature.One of these is the bifid median nerve.Due to its relatively higher cross-sectional area, it can facilitate compression of the median nerve in the carpal tunnel.Therefore, bifid median nerve is relatively common in patients with CTS.Some studies have shown that the bifid median nerve has an effect on surgical failure in the treatment of carpal tunnel syndrome.Apart from surgical treatment, perineural injection with corticosteroids is a treatment method that has been used for a long time in the treatment of mild and moderate carpal tunnel syndrome.It is controversial whether bifid median nerve has a negative effect on treatment effectiveness.When looking at the literature, there is no previous study on this subject.With the introduction of ultrasound into our daily practice, the frequency of ultrasound-guided perineural injections has increased.Ultrasound allowed us to see variations in the median nerve before injection.The aim of the study is to compare the effectiveness of steroid injection in patients with CTS with bifid median nerve and patients with CTS with non-variant median nerve.It is also to investigate whether this anatomical variation has a negative effect on the treatment.

DETAILED DESCRIPTION:
Our study was designed as a prospective, double-blind randomized controlled study.Patients with an electrophysiological diagnosis of moderate CTS who applied to Etlik City Hospital Physical Therapy outpatient clinic will be included in the study.There are no sensitive groups.The research period was determined as 1 year.Sample size was calculated using the statistical power analysis programme G Power 3.1.9.4 for windows.Based on the study by Walker FO,the minimum number of patients required to achieve a significant change of 20 mm in VAS assesment before and after treatment(with a 5% Type 1 and Type 2 margin of error, 80% working power and 95% confidence interval) was found to be 17(total 34 patients) for each group.Considering the possibility of 20% loss during the study,ıt was decided to include at least 20(total 40) patients for each group.Demographic and clinical characteristics of Patients who met the inclusion criteria and completed the 'Informed Volunteer Consent Forum' will be recorded.The general pain of the patients will be evaluated with Visual Analog Scala,The symptom severity and functional status of the patients will be evaluated with the Boston Carpal Tunnel Questionnaire,The patients' hand grip strength measurement will be evaluated with a dynamometer.The patient hand diagram will be marked according to the patient's sensory symptoms.Median nerve cross-sectional area will be measured at the pisiform level with ultrasound, Distal motor latency and sensory nerve conduction velocity will be recorded with EMG.Pre-injection baseline assessments of participants will be made by a blinded investigator. In all patients, the median nerve will be visualized with ultrasound with a 12 MHz linear probe at the scaphoid-pisiform level.Afterwards, perineural injection(2cc:1cc 2% lidocaine hidroclorid+1cc betamethasone) will be performed using an in-plane approach around the median nerve.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being clinically diagnosed with Carpal Tunnel Syndrome
* Confirmation of mild and moderate Carpal Tunnel Syndrome diagnosis with EMG
* Diagnosis of bifid median nerve after ultrasound evaluation, No variation was detected for the control group either.
* Having typical Carpal Tunnel Syndrome symptoms for at least 3 months

Exclusion Criteria:

* History of polyneuropathy, brachial plexopathy, thoracic outlet syndrome, or wrist surgery
* History of Inflammatory arthritis, hypothyroidism, pregnancy,rheumatological disorders or heart battery
* current warfarin use, Prior steroid injection for CTS, trauma or neoplasm at the injection site, hypersensitivity to corticosteroids or skin infection at the injection site
* other median nerve variations and presence of persistent median artery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-09-14 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) | This evaluation will be made and recorded at the baseline, at the 4th and 12th weeks after the procedure.
  Global pain:The VAS used for pain assessment consists of a line drawn in the form a ruler,and numbers from 0 to 10(with 0 as ''no pain'' and 10 as ''unbearable pain'' ) were asked to score.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | This evaluation will be made and recorded at the baseline, at the 4th and 12th weeks after the procedure.
  symptom severity and functional status scale
Electromyography | This evaluation will be made and recorded at the beginning.
  Distal motor latency and sensory nerve conduction velocity
Dynamometer | This evaluation will be made and recorded at the baseline, at the 4th and 12th weeks after the procedure
  Hand grip strength measurement test
Ultrasound | This evaluation will be made and recorded at the beginning.
  Median nerve cross-sectional area measurement at the pisiform level

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül Yaman, specialist, Study Chair — Ankara Etlik City Hospital; Başak Mansız Kaplan, assoc. prof, Study Chair — Ankara Etlik City Hospital; Aslıhan Uzunkulaoğlu, assoc. prof, Study Chair — Ankara Etlik City Hospital; Selin Çelebier, assistant dr, Study Chair — Seli̇n Çelebi̇er
Locations (1):
- Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayrak IK, Bayrak AO, Kale M, Turker H, Diren B. Bifid median nerve in patients with carpal tunnel syndrome. J Ultrasound Med. 2008 Aug;27(8):1129-36. doi: 10.7863/jum.2008.27.8.1129. PMID 18645070
- [Background] Theofilopoulou S, Katouni K, Papadopoulos V, Pappas N, Antonopoulos I, Giavopoulos P, Chrysikos D, Filippou D. Variations of the Median Nerve and Carpal Tunnel Syndrome: a Systematic Review of the Literature. Maedica (Bucur). 2023 Dec;18(4):699-704. doi: 10.26574/maedica.2023.18.4.699. PMID 38348062
- [Background] Granata G, Caliandro P, Pazzaglia C, Minciotti I, Russo G, Martinoli C, Padua L. Prevalence of bifid median nerve at wrist assessed through ultrasound. Neurol Sci. 2011 Aug;32(4):615-8. doi: 10.1007/s10072-011-0582-8. Epub 2011 Apr 30. PMID 21533564